CLINICAL TRIAL: NCT00905294
Title: ADAMTS-13 Activity, Von Willebrand Factor and Platelet-Monocyte Aggregation in Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Study of ADAMTS-13 Activity, Von Willebrand Factor and Platelet-Monocyte Aggregation in Coronary Artery Disease
Acronym: ADVANCE-PCI
Status: Terminated | Type: Observational
Why Stopped: Funding withdrawn
Sponsor: University College Cork (Other)
Collaborators: Royal College of Surgeons, Ireland (Other)
Responsible Party: Principal Investigator, Professor Noel Caplice, Professor, Cardiovascular Sciences, University College Cork
Other Study IDs: INFACTs 2009-001
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- coronary artery disease: Subjects with coronary artery disease undergoing percutaneous coronary intervention
  Interventions: Other: Blood draws

INTERVENTIONS:
Other: Blood draws — Observational: blood draws only

SUMMARY:
The purpose of this research is to determine the relationship between proteins and enzymes in the blood and how they work with platelets to form blood clots in patients with coronary artery disease. The investigators hypothesize that the relationship between these factors could potentially be useful in identifying patients at higher risk for heart attacks.

ELIGIBILITY:
Inclusion Criteria:

* Admission to hospital with suspected index event of Non-ST-Elevation Myocardial Infarction (NSTEMI), Unstable Angina (UA) or Stable Angina (SA)
* Planned percutaneous coronary intervention during admission

Exclusion Criteria:

* Recent history (< 6 months) of an acute coronary syndrome (other than current admission) or stroke
* Recent history (< 6 months) of major surgery, trauma or thromboembolic event
* Percutaneous coronary or peripheral intervention or any stent placement performed within the past 6 months
* Current evidence of infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease undergoing percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
relationships between ADAMTS-13 activity, von Willebrand factor antigen and platelet-monocyte aggregates levels | change from baseline to after percutaneous coronary intervention
  Assess the relationships between ADAMTS-13 activity, von Willebrand factor antigen and platelet-monocyte aggregates levels in subjects with coronary artery disease prior to and after undergoing PCI in this exploratory study

CONTACTS AND LOCATIONS:
Overall Officials: Noel M. Caplice, M.D, Ph.D., Principal Investigator — University College Cork, Ireland; Dermot Kenny, M.D., Study Director — Royal College Surgeons in Ireland; David Foley, M.B., Study Director — Beaumont Hospital, Dublin, Ireland
Locations (2):
- Ireland (2):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin